CLINICAL TRIAL: NCT04745091
Title: Complete Clinical Response With MRI Split Scar Sign as a Predictor to Complete Pathologic Response After Neoadjuvant Chemoradiation in Rectal Cancer
Brief Title: MRI Split Scar Sign as a Predictor to Complete Pathologic Response After Neoadjuvant Chemoradiation in Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Khaled Madbouly, Professor of Surgery, Alexandria University
Other Study IDs: 0201372
Record Dates: First submitted 2021-01-30; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Rectum Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — rectal cancer specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: total mesorectal excision — excision of the rectum with complete excision of the mesorectum

SUMMARY:
Patients with middle or low rectal cancer who receive neoadjuvant chemoradiation and achieve complete clinical response while their pelvic MRI have split scar sign are included. Patients will have total mesorectal excision and pathologic complete response will be assessed

DETAILED DESCRIPTION:
Patients with middle or low rectal cancer who have T3-4 and/ or N+ will be included. Patients will receive neoadjuvant chemoradiation in the form of pelvic irradiation by 50.4 thousands grays together with radio sensitization by 5-FU or oxaliplatin, 8 months after completion of neoadjuvant chemoradiation patients will be assessed clinically and radiologically. Complete clinical response is diagnosed if clinically no tumor is felt or just small scar and no tumor appears in MRI. Of these patients who achieve complete clinical response we will pick up cases who have split scar sign in the pelvic MRI. Patients will have total mesorectal excision 8-11 weeks after completion of neoadjuvant chemoradiation and pathologic complete response will be assessed. Correlation will be done between preoperative clinical response and postoperative pathologic response

ELIGIBILITY:
Inclusion Criteria:

middle and low rectal cancer

Exclusion Criteria:

* Distant metastasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: locally advance middle and low rectal cancer
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete pathologic response | after surgical excision with follow up of an average of 1 year
  disappearance of tumor from resected specimen

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Madbouly, MD, PhD, Principal Investigator — University of Alexandria

IPD SHARING:
Plan to Share IPD: Undecided
no approval yet from ethical committee to share data. Not written in patients' consent yet